CLINICAL TRIAL: NCT02117362
Title: Phase IB Study of a Galectin Inhibitor (GR-MD-02) and Ipilimumab in Patients With Metastatic Melanoma
Brief Title: Galectin Inhibitor (GR-MD-02) and Ipilimumab in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other); Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-004A
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Ipilimumab; Yervoy; Galectin; GR-MD-02; galactoarabino-rhamnogalacturonate; galectin-3 inhibitor; Providence Health & Services; Earle A. Chiles Research Institute; Robert W. Franz Cancer Center; Immunotherapy
MeSH Terms: conditions — Melanoma | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 1 mg/kg GR-MD-02 administered 1 hour before 3 mg/kg of ipilimumab on Days 1, 22, 43, and 65.
  Interventions: Biological: 1 mg/kg GR-MD-02; Biological: Ipilimumab
- Cohort 2 (Experimental): 2 mg/kg GR-MD-02 administered 1 hour before 3 mg/kg of ipilimumab on Days 1, 22, 43, and 65.
  Interventions: Biological: 2 mg/kg GR-MD-02; Biological: Ipilimumab
- Cohort 3 (Experimental): 4 mg/kg GR-MD-02 administered 1 hour before 3 mg/kg of ipilimumab on Days 1, 22, 43, and 65.
  Interventions: Biological: 4 mg/kg GR-MD-02; Biological: Ipilimumab
- Cohort 4 (Experimental): 8 mg/kg GR-MD-02 administered 1 hour before 3 mg/kg of ipilimumab on Days 1, 22, 43, and 65.
  Interventions: Biological: 8 mg/kg GR-MD-02; Biological: Ipilimumab

INTERVENTIONS:
Biological: 1 mg/kg GR-MD-02 — 1 mg/kg GR-MD-02 on Days 1, 22, 43, and 65.
  Other Names: galectin-3 inhibitor; galactoarabino-rhamnogalacturonate
  Arms: Cohort 1
Biological: 2 mg/kg GR-MD-02 — 2 mg/kg GR-MD-02 on Days 1, 22, 43, and 65.
  Other Names: galectin-3 inhibitor; galactoarabino-rhamnogalacturonate
  Arms: Cohort 2
Biological: 4 mg/kg GR-MD-02 — 4 mg/kg GR-MD-02 on Days 1, 22, 43, and 65
  Other Names: galectin-3 inhibitor; galactoarabino-rhamnogalacturonate
  Arms: Cohort 3
Biological: 8 mg/kg GR-MD-02 — 8 mg/mg GR-MD-02
  Other Names: galectin-3 inhibitor; galactoarabino-rhamnogalacturonate
  Arms: Cohort 4
Biological: Ipilimumab — 3 mg/kg ipilimumab on Days 1, 22, 43, and 65
  Other Names: Yervoy; Anti-CTLA 4

SUMMARY:
The goal of this study is to determine a safe dose of GR-MD-02 used in combination with the FDA-approved dose of ipilimumab (3 mg/kg) in patients who have advanced melanoma. GR-MD-02 is a galectin. Galectins are a family of proteins that have numerous functions in normal mammalian biology including the facilitation of cell-cell interactions, regulation of cell-death and regulation of immune system responses. The hypothesis is that a safe dose of GR-MD-02 when given with the FDA-approved dose of ipilimumab can be found.

DETAILED DESCRIPTION:
This study will employ a 3+3 phase I design with dose escalation of GR-MD-02 in conjunction with the standard therapeutic dose of ipilimumab in patients with advanced melanoma for whom ipilimumab would be considered standard of care. In addition to monitoring for toxicity and clinical response, blood samples will be obtained to assess immunologic measures relevant to galectin biology and ipilimumab T-cell check-point inhibition

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or unresectable melanoma for whom treatment with ipilimumab is indicated. Histological confirmation of melanoma will be required by previous biopsy or cytology.
* Patients must be ≥ 18 years of age.
* Eastern Collaborative Oncology Group (ECOG) performance status of 0-1.
* Women of childbearing potential must have a serum or urine pregnancy test performed within 72 hours prior to the start of protocol treatment. The results of this test must be negative in order for the patient to be eligible. In addition, women of childbearing potential as well as male patients must agree to take appropriate precautions to avoid pregnancy.
* No active bleeding.
* Anticipated lifespan greater than 12 weeks.
* Patients must sign a study-specific consent document.

Exclusion Criteria:

* Patients who have previously received a galectin antagonist
* Prior ipilimumab to treat metastatic melanoma (prior ipilimumab in the adjuvant setting is permitted if the patient did not experience ≥ grade 3 toxicity related to immunotherapy.
* Patients with active autoimmune disease except for autoimmune thyroiditis or vitiligo.
* Patients with history of colitis
* Patients with untreated brain metastases. Patients with treated brain metastases who demonstrate control of brain metastases with follow-up imaging 4 or more weeks after initial therapy are eligible.
* Other active metastatic cancer requiring treatment.
* Patients with active infection requiring antibiotics.
* Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus.
* Laboratory exclusions (to be performed within 28 days of enrollment):
* Need for chronic steroids. Inhaled corticosteroids are acceptable.
* Inability to give informed consent and comply with the protocol. Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.
* Any medical condition that in the opinion of the Principal Investigator would compromise the safety or conduct of the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05-08 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
Determine a safe dose of GR-MD-02 used in combination with the approved dose of ipilimumab (3 mg/kg) | 21 Days
  Patients return to clinic 9 times in 85 days, receiving treatment on Days 1, 22, 43, and 65. Patients will have physical exams, blood tests, and toxicity evaluations by a research nurse during this time to identify any protocol-defined dose limiting toxicity.

SECONDARY OUTCOMES:
Response rate to combined therapy | 85 Days
  Tumor burden assessments will occur at screening, Day 85, and every 12 weeks thereafter to determine the response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Curti, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Providence Cancer Center — http://oregon.providence.org/our-services/p/providence-cancer-center/